CLINICAL TRIAL: NCT02238301
Title: Study of the Fetoplacental BOLD Effect in Pregnant Women Using Functional MRI
Brief Title: Evaluation of Fetoplacental Oxygenation With Functional MRI in Pregnant Women
Acronym: BOLD-FP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P130924
Record Dates: First submitted 2014-09-09; First posted 2014-09-12 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Intrauterine Growth Restriction
Keywords: Intrauterine growth restriction; BOLD effect
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients "test" (pregnant women with a eutrophic fetus) (Other): Test the type of mask, oxygen flow and duration of oxygenation, adjustment of MRI machine Adjustment of MRI machine (choice of antenna calibration, verifying Settings of each sequence, adaptation of the number of cuts for the duration of each sequence, checking the correct execution of the succession of sequences, settings of total examination time)
  Interventions: Other: Bold sequence patients test
- Pregnant women with a diagnosis of IUGR fetuses (Active Comparator): Measure of the BOLD effect in the feto-placental units of IUGR fetuses
  Interventions: Other: Bold + ASL sequence
- Pregnant women with eutrophic fetuses (Active Comparator): Measure of BOLD effects of fetal-placental unit eutrophic fetuses
  Interventions: Other: Bold + ASL sequence

INTERVENTIONS:
Other: Bold sequence patients test — Develop the hyperventilation protocol (speed, duration ...) and the choice of type of mask oxygenation better tolerated by patients. Sequences beginning with a low oxygen flow (2L/mn) then progressively increasing to obtain the BOLD effect required
  Arms: Patients "test" (pregnant women with a eutrophic fetus)
Other: Bold + ASL sequence — A first sequence BOLD+ASL will be launched in ambient air. The second sequence is repeated BOLD 5 minutes after power maternal hyperventilation.
  Sequences will focus on the fetus and placenta but will also include maternal liver to validate maternal hyperoxygenation.
  Arms: Pregnant women with a diagnosis of IUGR fetuses; Pregnant women with eutrophic fetuses

SUMMARY:
The purpose of this study is to evaluate the use of functional MRI in pregnant women as a non-invasive diagnostic tool to detect placental insufficiency and differentiate healthy fetuses from the intra-uterine growth restricted ones. Functional MRI in pregnant women can detect a variation of the MRI signal (called BOLD effect) from the placenta and the fetus when the mother is breathing pure oxygen. This study aims hence to demonstrate the difference in the BOLD effect between normal feto-placental units and growth restricted ones.

DETAILED DESCRIPTION:
Intrauterine growth restriction (IUGR) is associated with important maternal and perinatal morbidity and mortality. IUGR is typically secondary to defective oxygenation, leading to placental insufficiency.

Measurements made in the umbilical cord after puncture fetal blood showed that compared to normal fetuses, fetuses with IUGR are often hypoxic, hypercapnic and acidotic. Pathological placental and fetal oxygenation is considered as a main element of IUGR. To this day, there is no non-invasive exploration method of this oxygenation. The only ways to monitor IUGR are "indirect" ultrasonic analysis of fetal growth and uteroplacental Doppler spectra. Functional BOLD (Blood Oxygen Level dependent) MRI, already used to investigate cerebral, tumor, cardiac oxygenation, highlights local variations of oxygenation. The purpose of this study is to obtain non invasive data of fetoplacental oxygenation through functional BOLD MRI. Comparing data on eutrophic fetuses and IUGR fetuses will determine the potential contribution of this technique in the diagnosis, treatment and medical management of dysfunctional placentas associated with an increased risk of IUGR.

a fetal MRI in the pediatric radiology department of Necker-Enfants Malades Hospital or Robert Debré Hospital, for fetal or placental indications as part of usual workup, will be invited to participate in this protocol. At the waning of the scheduled fetal MRI, patients will subsequently receive an additional BOLD and ASL sequence before and after maternal hyperoxygenation.

Patients will be included in three centers : Necker Hospital, Robert Debré Hospital and Louis Mourier Hospital. Only at Necker Hospital: a subgroup of patients will be included at the beginning of the protocol for the adjustment of the settings of the MRI machine, for the determination of BOLD sequences' parameters, as well as the selection of the most adapted type of oxygenation mask.

In the three centers, investigators will include patients with IUGR fetuses and patients with a eutrophic fetus.

A total of two visits (selection visit and baseline) are scheduled for all patients in this trial. Patient selection will be done during a ultrasound visit. Patients can give their consent on the same day or on the MRI appointment day; in all cases the consent will be signed on the day of the appointment MRI.

The flow and duration of the oxygenation of the initial group "test patients" will be determined before completion of the examination; for other patients, the flow rate will be determined based on the results of this first group.

The duration of the BOLD sequence will be around 10 minutes. The sequences will focus on the feto-placental unit.

A first BOLD sequence will be launched under ambient air. The second BOLD sequence will be repeated after 5 minutes of maternal hyperoxygenation.

MRI data will be saved and analyzed at the Laboratory of Imaging Research of the team 2 of Paris Cardiovascular Research Center (INSERM U970).

The data necessary for the statistical analysis of the study are collected from the medical file of patients included in the study. Data entry will be performed by a research technician on electronic media via an internet browser.

The inclusion period will be of 57 months. Each woman's duration of participation will be 1 hour. The maximum duration of the study will be 57 months.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient with a singleton pregnancy
* Patient between 18 and 37 gestational weeks
* Informed consent signed by the patient
* Patient affiliated to a social security scheme (beneficiary or assignee) Specific criteria for patients with a eutrophic fetus
* Patient with fetal eutrophic on sonographic fetal weight estimation Specific criteria for patients with an IUGR-fetus Patient with a fetus presenting intra-uterine growth restriction diagnosed by ultrasound (<5th percentile).

Exclusion Criteria:

* Patient with the usual contra-indications for MRI
* Patient with an abdominal circumference> 125 cm
* Patient with a multiple pregnancy
* Patient with placenta accreta or percreta
* Patient with a pregnancy after long history of infertility and medically assisted procreation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-02-18 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Highlight a placental BOLD effect | at inclusion
  Measured as the difference between the T2* of the placenta under the ambient air and under hyperoxygenation.

SECONDARY OUTCOMES:
Number of patients with positive difference of signal intensity of maternal liver, under the ambient air and under hyperoxygenation | at inclusion
BOLD effect in the fetal liver and brain of eutrophic fetuses | at inclusion
  Measure the BOLD effect in the fetal liver and brain of eutrophic fetuses
BOLD effect in the fetal liver and brain of IUGR fetuses | at inclusion
  Measure the BOLD effect in the fetal liver and brain of IUGR fetuses
BOLD effect in the maternal liver of IUGR fetuses | at inclusion
  Measure a Bold effect in the maternal liver of IUGR fetuses
Measure a Bold effect in the placenta of IUGR fetuses | at inclusion
Feasibility : number of possible perfusion measure | at inclusion
Feasibility : percent of possible perfusion measure | at inclusion
Compare the placental perfusion between eutrophic and RCIU fetuses | at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Laurent SALOMON, MD, PhD, Study Director — Hospital Necker - Enfants Malades - Public Hospitals of Paris
Locations (1):
- Necker - Enfants Malades Hospital (Assistance Publique des Hopitaux de Paris), Paris, France

REFERENCES:
- [Background] Jacquier M, Chalouhi G, Marquant F, Bussieres L, Grevent D, Picone O, Mandelbrot L, Mahallati H, Briand N, Elie C, Siauve N, Salomon LJ. Placental T2* and BOLD effect in response to hyperoxia in normal and growth-restricted pregnancies: multicenter cohort study. Ultrasound Obstet Gynecol. 2024 Apr;63(4):472-480. doi: 10.1002/uog.27496. PMID 37743665